CLINICAL TRIAL: NCT06756542
Title: Utilizing Large Language Models to Augment Family Conversations in the Intensive Care Unit
Brief Title: Evaluating the Use of Artificial Intelligence to Improve Family Conversations for Intensive Care Patients and Their Families
Status: Recruiting | Type: Observational
Sponsor: Davy van de Sande (Other)
Responsible Party: Sponsor-Investigator, Davy van de Sande, Coordinating Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2024-0733
Record Dates: First submitted 2024-12-02; First posted 2025-01-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care Medicine; Critical Care
Keywords: intensive care; artificial intelligence; large language models; administration reduction; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study looks at how artificial intelligence (AI), like generative pre-trained transformer (GPT-4), can help doctors in the intensive care unit (ICU) save time and improve communication with families. Right now, doctors spend a lot of time writing notes after family conversations, which takes time away from patient care. The investigators are testing whether AI can create accurate and easy-to-understand summaries of these conversations, making it quicker for doctors to document and clearer for families to understand. ICU doctors and adult family members of patients will take part in this study, with their full consent. The goal is to see if this new technology can make life easier for doctors while helping families better understand medical information.

ELIGIBILITY:
Inclusion Criteria:

* Informed-consent is signed by all participating family members during the conversation.
* Informed-consent is signed by the ICU healthcare professionals.
* The patient of the family must be admitted to the adult ICU.
* All participating family members must be 18 years or older.
* The family conversation must be in Dutch.

Exclusion Criteria:

* Trained to interpret medical jargon and/or intensive care terminology specifically
* Difficulty reading and/or writing in the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care professionals performing formal family conversations and family members of patients admitted to the adult intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Documentation quality of family conversations | Within 30 days after the family conversation.
  The primary outcome measure is the documentation quality of family conversations, evaluated using a modified Physician Documentation Quality Instrument-9. Originally validated for progress notes and discharge summaries, Physician Documentation Quality Instrument-9 scores notes on nine attributes (accurate, thorough, useful, organized, comprehensible, succinct, synthesized, consistent, up-to-date) using a 1-5 scale (1 = "not at all," 5 = "extremely"), for a total ranging from 9 to 45. To adapt it for AI-generated text, the investigators removed the "up-to-date" domain (focused on whether the note includes the latest test results/recommendations) and added two new attributes: freedom from hallucinations (unfounded information) and freedom from bias (discriminatory data, algorithms, or heuristics). These additions address potential pitfalls in large language model outputs, such as introducing incorrect content or skewed results.

SECONDARY OUTCOMES:
Time spent on documentation by ICU clinicians | Within one day after the family conversation.
  The time clinicians spend on post-conversation documentation will be measured for both traditional and ambient listening methods. This outcome aims to quantify the efficiency of the ambient listening technology in reducing administrative burden.
Family satisfaction | Within 30 days after the family conversation.
  Family members' feedback on their satisfaction with the intensive care unit (ICU) communication process. Satisfaction will be measured using a structured questionnaire administered after reviewing a simplified ambient-generated note. The survey includes 16 questions: 5 about demographics (age, education, occupation, and reading skills); 3 adapted from the validated Family Satisfaction with the ICU-24 survey (score range: 1-5, higher scores indicate greater satisfaction) to assess clarity, completeness, and overall satisfaction; and 10 evaluating the summary's readability and utility at a B1 language proficiency level.

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Gommers, MD PhD, Study Director — Intensive Care Adults, Erasmus University Medical Center, Rotterdam, the Netherlands; Michel E. van Genderen, MD PhD, Principal Investigator — Intensive Care Adults, Erasmus University Medical Center, Rotterdam, the Netherlands
Locations (2):
- Netherlands (2):
  - Erasmus University Medical Center, Rotterdam, South Holland
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided